CLINICAL TRIAL: NCT01410071
Title: Evaluation of Gastrointestinal Symptoms and Quality of Life in Patients With Sphincter of Oddi Dysfunction: Evaluation of the Differences Between Those Undergoing Endoscopic Therapy vs.Conservative Care
Brief Title: Evaluation of Gastrointestinal Symptoms and Quality of Life in Patients With Sphincter of Oddi Dysfunction
Status: Terminated | Type: Observational
Why Stopped: Analysis of designed comparison groups not viable
Sponsor: Wisconsin Center for Advanced Research (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Nalini Guda MD, Wisconsin Center for Advanced Research, Division of GI Associates LLC
Other Study IDs: S-05-130E
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Sphincter of Oddi Dysfunction; Abdominal Pain
Keywords: Sphincter of Oddi Dysfunction
MeSH Terms: conditions — Sphincter of Oddi Dysfunction; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sphincter of oddi dysfunction: endoscopic therapy vs conservative care

SUMMARY:
The purpose of this research study is to see if there is a significant difference in improvement of symptoms and quality of life of those undergoing endoscopic therapy versus those wanting to control their symptoms with medicines or those who just want to wait and watch.

DETAILED DESCRIPTION:
Sphincter of Oddi is a complex muscular structure which regulates the biliary and pancreatic outflow into the duodenum. Resting pressures >40mm of Hg are considered abnormal. Individuals with elevated resting/basal biliary or pancreatic sphincter pressures are thought to have sphincter of oddi dysfunction. Sphincter dysfunction often manifests as pain and the nature of the pain is dependent on the involvement of either the biliary or the pancreatic sphincter. In most instances the pain is debilitating and could impair the quality of life. Endoscopic therapy- either biliary or pancreatic sphincterotomy, is often performed for relief of symptoms. Data regarding the efficacy of such an approach are limited. A recent systematic review by the Cochrane reviewers has found only two randomized controlled trials evaluating the efficacy of sphincterotomy for relief of symptoms in those with sphincter of Oddi dysfunction and there were no data evaluating the quality of life or the health economics of such an approach.

ELIGIBILITY:
Inclusion Criteria:

* over age 18
* suspected history and clinical features suggestive of sphincter of oddi dysfunction

Exclusion Criteria:

* prior history of endoscopic therapy for sphincter of oddi dysfunction
* no proven sphincter of oddi dysfunction on manometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: physician's private practice/clinic patients presenting with suspected sphincter of oddi dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
symptom improvement | one year

SECONDARY OUTCOMES:
improved quality of life | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nalini M Guda, MD, Principal Investigator — GI Associates
Locations (1):
- Wisconsin Center for Advanced Research, Milwaukee, Wisconsin, United States